CLINICAL TRIAL: NCT02720926
Title: A Phase 1 Study of TKI 258 in Combination With Xeloda and Oxaliplatin in Upfront Treatment of Advanced Colorectal and Gastric Cancer With a Dose Expansion Cohort in Advanced Gastric Cancer
Brief Title: Study of TKI 258 in Combination With Xeloda and Oxaliplatin in Advanced Colorectal and Gastric Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unafavourable toxicity profile
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC 10-03
Record Dates: First submitted 2012-05-14; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer; Gastric Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 combined with Xeloda/Oxaliplatin (Experimental): TKI258 200 mg once a day (OD) 5 days on/2 days off Capecitabine (Xeloda) 2000 mg/m2 bid d1-14 Oxaliplatin 130mg/m2 d1 q21days
  Interventions: Drug: Xeloda,; Drug: Oxaliplatin; Drug: TKI258

INTERVENTIONS:
Drug: Xeloda, — Capecitabine (xeloda): 2000mg/m2, twice a day on Day 1-14;
  Other Names: capecitabine
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 day 1 every 21days
Drug: TKI258 — 4 dose levels of TKI258: 200mg, 300mg, 400mg, 500mg once daily, 5days on and 2 days off;

SUMMARY:
Standard "3+3" dose escalation design of TKI258/XELOX in advanced gastric/gastro-oesophageal and colorectal cancer.

DETAILED DESCRIPTION:
This is a "3+3" dose escalation design with 4 pre-defined TKI258 dose levels (200mg, 300mg, 400mg and 500mg daily with 5 days on and 2 days off schedule) in combination with a fixed standard dose of XELOX (Capecitabine and Oxaliplatin) to establish the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed gastric, gastro-oesophageal or colorectal adenocarcinoma.
2. The gastric or gastro-oesophageal cancer must be locally advanced unresectable or metastatic. Colorectal cancer must be metastatic and for which subsequent resection of all metastatic disease is assessed not to be feasible.
3. Age >18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%, see Appendix A).
5. Life expectancy of greater than 3 months
6. Patients must have normal organ and marrow function as defined below:

   * leukocytes >3,000/mcL
   * absolute neutrophil count >1,500/microliter (mcL) TKI258/XELOX phase 1 protocol version 3.3 Dated 30 November 2011 1 3
   * platelets >100,000/mcL
   * total bilirubin <= 1.5 x upper limit of normal (ULN)
   * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits OR
   * creatinine clearance >55 mL/min for patients with creatinine levels above institutional normal.
7. The effects of TKI258 and XELOX on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Baseline left ventricular ejection fraction (LVEF) >= 50%
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients are not considered to have a "currently active" malignancy if they have TKI258/XELOX phase 1 protocol version 3.3 Dated 30 November 2011 1 4 completed therapy and are considered to have a less than 30% risk of relapse.
2. Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TKI258 or XELOX, breastfeeding should be discontinued if the mother is treated with TKI258 or XELOX.
3. Patients with prior history of transient ischemia attack or cerebrovascular disease or prior history of ischemia heart disease or myocardia infarction and 2 or more risk factors: ever smoker with > 30 packs per year exposure or on medication for diabetes mellitus or hypertension or hyperlipidemia.
4. In addition for the Beginning at dose expansion cohort, the following exclusion criteria apply:

   * Patients who are not agreeable for collection of tumor tissue for correlative studies
   * Patients from whom tumor tissue for correlative studies cannot be safely obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determine the recommended phase 2 dose of TKI258 in combination with XELOX (Capecitabine and Oxaliplatin) | 42 days

SECONDARY OUTCOMES:
Describe the toxic effects of TKI258 when administered in combination with XELOX chemotherapy. | one year
  Toxicity will be graded using CTCAE version 4.0
Measure the Area under the plasma concentration versus time curve (AUC) of TKI258 at specific timepoints | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Iain BH Tan, Dr, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No